CLINICAL TRIAL: NCT00941460
Title: Dose-intensified Rechallenge With Temozolomide, One Week On One Week Off Versus Three Weeks On One Week Off in Patients With Progressive or Recurrent Glioblastoma
Brief Title: Comparison of Two Dosing Regimens of Temozolomide in Patients With Progressive or Recurrent Glioblastoma
Acronym: DIRECTOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Dr. Wolfgang Wick (Other)
Collaborators: Essex Pharma GmbH (Industry)
Responsible Party: Sponsor-Investigator, Prof. Dr. Wolfgang Wick, Coordinating Investigator, Heidelberg University
Organization: Heidelberg University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIRECTOR; 2008-006871-60 (EudraCT Number); ISRCTN68738654 (Registry Identifier: controlled-trials)
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Glioblastoma
Keywords: progressive or recurrent glioblastoma; temozolomide; dose intensification; comparison of two dosing regimens
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- one week on one week off (Experimental): One week on temozolomide is followed by a week without temozolomide.
  Interventions: Drug: Temozolomide in both arms
- three weeks on, one week off (Experimental): Temozolomide is given over 3 weeks, followed by a week without temozolomide.
  Interventions: Drug: Temozolomide in both arms

INTERVENTIONS:
Drug: Temozolomide in both arms — initial dose 120 mg/m2 in arm A
  Other Names: Temodal
  Arms: one week on one week off
Drug: Temozolomide in both arms — initial dose 80 mg/m2 in arm B
  Other Names: Temodal
  Arms: three weeks on, one week off

SUMMARY:
For patients with progressive or recurrent glioblastoma there is no standard therapy. One strategy is re-exposure to temozolomide in a higher dose. This increase in dosing can be done by 2 regimens. Aim of this study is to compare these 2 dosing regimens concerning toxicity. In study arm A patients receive temozolomide for one week, followed by a week without temozolomide. In study arm B patients receive temozolomide for three weeks, followed by a week without temozolomide. The regimen that is less toxic will be selected for further evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Progressive or recurrent glioblastoma documented by MRI no earlier than 180 days after first surgery for glioblastoma and no earlier than 90 days after completion of radiotherapy.
* Histological diagnosis of glioblastoma
* Tissue available for the determination of MGMT promoter methylation in the primary tumor or from the recurrent tumor if a patient undergoes a surgical procedure at recurrence prior to study entry.
* Prior treatment with temozolomide administered concomitantly with radiotherapy and at least for two cycles (5/28) as an adjuvant treatment
* Informed consent
* Age 18-80 years
* Karnofsky performance score > 50%
* Neutrophil counts > 1 500/µl
* Platelet counts > 100 000/µl
* Hemoglobin > 10 g/dl
* Serum creatinin < 1.5-fold upper normal range
* ASAT or ALAT < 3-fold upper normal range unless attributed to anticonvulsants
* Alkaline phosphatase < 3-fold upper normal range
* Women with childbearing potential must have a negative serum pregnancy test ≤14 days prior to study enrollment
* Willingness to apply contraception according to local requirements (as stated in patient information)

Exclusion Criteria:

* Progressive or recurrent glioblastoma documented by MRI earlier than 180 days after first surgery for glioblastoma and earlier than 90 days after completion of radiotherapy.
* Treatment with any chemotherapy other than temozolomide according to the schedule of the EORTC NCIC trial (Stupp et al. N Engl J Med 2005;352:987-996) except that an adjuvant starting dose of 200 mg/m2 and more than 6 cycles of adjuvant temozolomide are allowed
* Prior systemic or local treatment with DNA-damaging agents, tyrosine kinase inhibitors or anti-angiogenic agents for any cancer
* Allergy to or other intolerability of temozolomide
* Unable to undergo MRI
* Past medical history of diseases with poor prognosis, e.g. severe coronary heart disease, severe diabetes, immune deficiency, residual deficits after stroke, severe mental retardation
* HIV infection
* Pregnancy
* Breast feeding
* Treatment within in any other clinical trial parallel to the treatment phase of the current study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2009-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Median time to treatment failure. Treatment failure is reached (i) upon tumor progression as outlined in protocol (ii) if treatment has to be terminated due to toxicity or (iii) if the patient dies for any reason. | up to one year

SECONDARY OUTCOMES:
progression free survival | up to two years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Weller, Prof. Dr., Study Chair — University of Zurich
Locations (16):
- Austria (2):
  - Landesnervenklinik Wagner-Jauregg, Linz
  - Medical University Vienna, Department of Internal Medicine I, Vienna
- Germany (12):
  - Charite, Department of Neurosurgery, Berlin
  - Knappschaftskrankenhaus, Department of Neurology, Bochum
  - University Hospital Bonn, Department of Neurology, Bonn
  - Klinik für Allgemeine Neurochirurgie, Cologne
  - University Hospital Düsseldorf, Düsseldorf
  - Klinikum der Johann-Wolfgang von Goethe-Universität, Dr. Senckenbergisches Institut für Neuroonkologie, Zentrum für Neurologie und Neurochirurgie, Frankfurt
  - University Hospital Freiburg, Freiburg im Breisgau
  - University Hospital Heidelberg, Department of Neurooncology, Heidelberg
  - Saarland University, Department of Neurosurgery, Homburg/ Saar
  - Klinik und Poliklinik für Neurochirurgie, Leipzig
  - Ludwig Maximilians University of Munich , Grosshadern Hospital, Department of Neurosurgery, Munich
  - University of Regensburg, Department of Neurology, Regensburg
- Switzerland (2):
  - University Hospital Zurich, Department of Neurology, Zurich, CH
  - Centre Hospitalier Universitaire Vaudois and University of Lausanne, Lausanne